CLINICAL TRIAL: NCT05466500
Title: The Efficacy of Intravenous Dexamethasone on the Duration of Analgesia of Ultrasound Guided Axillary Brachial Plexus Block in Pediatric Patients Undergoing Below Elbow Orthopaedic Surgeries: A Randomized Control Trial
Brief Title: The Efficacy of Intravenous Dexamethasone on the Duration of Analgesia of Ultrasound Guided Axillary Brachial Plexus Block in Pediatric Patients Undergoing Below Elbow Orthopaedic Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed nabih youssef, Lecturer of anesthesia, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: N-53-2022
Record Dates: First submitted 2022-07-17; First posted 2022-07-20 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Axillary Brachial Plexus Block
MeSH Terms: interventions — Dexamethasone; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be done by computer generated numbers and concealed by serially numbered,opaque and sealed envelopes. The details of the series will be unknown to the investigators and the group assignment will be kept in asset of sealed envelopes each bearing only the case number on the outside. Prior to surgery the appropriate numbered envelopes will be opened by the nurse, the card inside will determine the patient group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound guided axillary block with intravenous dexamethasone (Active Comparator): The probe will be placed parallel to the anterior axillary fold at the axilla to identify the axillary artery and to identify the hyperechoic median, ulnar, and radial nerves in relation to the axillary artery. The musculocutaneous nerve which supplies the skin of the lateral side of the forearm had to be blocked also. It is found between the biceps brachii and coracobrachialis muscles .The needle is inserted in-plane from the anterior aspect and directed toward the posterior aspect of the axillary artery. All four nerves in the axillary region will be blocked and use of intravenous dexamethasone as an adjuvant to bupivacaine for Post-operative analgesia following sensory blockade of the axillary brachial plexus in paediatrics undergoing below elbow orthopaedic surgeries.
  Interventions: Procedure: Ultrasound guided axillary block with intravenous dexamethasone
- Ultrasound guided axillary block (Placebo Comparator): The probe will be placed parallel to the anterior axillary fold at the axilla to identify the axillary artery and to identifythe hyperechoic median, ulnar, and radial nervesin relation to the axillary artery. The musculocutaneous nerve which supplies the skin of the lateral side of the forearm had to be blocked also. It is found between the biceps brachii and coracobrachialis muscles .The needle is inserted in-plane from the anterior aspect and directed toward the posterior aspect of the axillary artery. All four nerves in the axillary region will be blocked
  Interventions: Procedure: Ultrasound guided axillary block

INTERVENTIONS:
Procedure: Ultrasound guided axillary block with intravenous dexamethasone — it will be given by one researcher using 2 mg/kg of 0.25% bupivacaine plus 0.1mg/kg dexamethasone intravenous
  Other Names: peripheral nerve block with dexamethasone; bupivacaine and dexamethasone intravenous
  Arms: Ultrasound guided axillary block with intravenous dexamethasone
Procedure: Ultrasound guided axillary block — it will be given by one researcher using 2 mg/kg of 0.25% bupivacaine
  Other Names: peripheral nerve block; bupivacaine only
  Arms: Ultrasound guided axillary block

SUMMARY:
Postoperative pain is a common manifestation in orthopedic patients, mainly due to intraoperative tissue damage , inadequate intraoperative pain assessment and management.

Axillary nerve block provides motor and sensory block with the distribution of the median, radial, ulnar and musculocutaneous branches so it can be conducted with upper limb orthopedic surgery in hand, rest and elbow surgery distal to the cubital fossa.Sensory blockade of the brachial plexus for perioperative analgesia leads to stable haemodynamics intraoperatively, smoother emergence from general anaesthesia and decreased need for supplemental analgesics or suppositories in the Post-operative period Intravenous (IV) dexamethasone has been used as an additive to local anesthetic for peripheral nerve blocks (PNBs) in adults with variable efficacy.To the best of our knowledge the efficacy of intravenous dexamethasone as adjuvant to bupivacaine in ultrasound guided axillary brachial plexus block in pediatrics has not been investigated

In this study the investigators will assess the analgesic effect of adding intravenous dexamethasone to bupivacaine in ultrasound guided axillary block in children undergoing upper limb orthopedic surgeries.

Objectives:

* To determine the effect of adding intravenous dexamethasone on the duration of analgesia .
* To determine the effect of adding intravenousdexamethasone on quality of analgesia

DETAILED DESCRIPTION:
This a randomized control trial is designed to include (60) patients ASA physical statusI-II patients ranging from(4) to(14)years old scheduled for upper limb orthopaedic surgery in the hand, wrist, and elbow distal to the cubital fossa.

Patients meeting the inclusion criteria will be randomly assigned to receive either :

Group A :Axillary block with 2 mg/kg of 0.25% bupivacaine. (n=30) Group B: Axillary block with 2 mg/kg of 0.25% bupivacaine plus 0.1mg/kg dexamethasone intravenous:(n=30)

All children will be anaesthetized in accordance with the local policy of the Abu El-Reesh pediatric hospital-Cairo university's pediatric anaesthetic unit. Except for oral clear liquids intake 2 hours before surgery, all children will fast for 6 hours. Patients will attend in the preparation room one hour before the operation to get a preoperative checkup, as well as their age and body weight will be recorded. Pre medicated by intramuscular injection of atropine 0.02 mg/Kg and midazolam 0.2 mg/Kg before insertion of intravenous (I.V) cannula.On arriving the operating room, heart rate (HR) ,oxygen saturation and non-invasive blood pressure will be continuously recorded, using standard monitor (Dräger infinity vista XL).

All patients will be induced with propofol 2 mg / kg , atracurium 0.5mg/kg and fentanyl 1μg/kg, then the patients will be intubated by appropriate size of endotracheal tube volume control ventilation (VCV) 5-7 ml/kg and respiratory rate will be adjusted to keep and PaCO2 levels between 30-35 mmHg using (G.E-Datex-Ohmeda, Avance CS2, USA) anesthesia machine. Anesthesia will be maintained with isoflurane 1 MAC with 50% oxygen in air, with the goal of keeping the BIS measurement between (40-60), and atracurium top-ups of 0.1mg/kg will be given every 30 minutes for neuromuscular blockade.Then the block will be conducted after general anesthesia by an expert anesthesiologist who is different from the anesthesiologist who provided anesthesia to the patient.

Axillary block

Axillary nerve block will be induced with patient in supine under GA with ultrasound SonoSite M Turbo (USA), the scanning probe will be the linear multi-frequency 6-13 MHz transducer (L25 x 6-13 MHz linear array).The probe will be protected with sterile cover, antiseptic betadine will be applied to the site of block injection , the operating arm will be abducted by 70 externally rotated, and the elbow will be flexed to ~90. Within the axillary crease the probe position will be placed sagittal where bounded by the pectoralis major antero-medially and the latissimus dorsi and teres major posteromedial.

The probe will be placed parallel to the anterior axillary fold at the axilla to identify the axillary artery and to identify the hyperechoic median, ulnar, and radial nerves in relation to the axillary artery. The musculocutaneous nerve which supplies the skin of the lateral side of the forearm had to be blocked also. It is found between the biceps brachii and coracobrachialis muscles .The needle is inserted in-plane from the anterior aspect and directed toward the posterior aspect of the axillary artery. All four nerves in the axillary region will be blocked. The block will be applied by 50-mm block needle 22 gauge at cephalic side of the probe. The same volume of local anesthetic will be used in each group with 2 mg/kg of 0.25% bupivacaine. Group A will receive 2ml of saline solution i.v after completing the block,Group B will receive 0.1mg/kg dexamethasone i.v after completing the block.

The time passed between the entrance of the needle into the skin and the injection's completion is referred to as axillary block performance time.The end of the local anesthetic solution injection will be considered the time zero to assess the blockade effectiveness. The surgical procedure will be start after 15-20 min.

If there is an increase in heart rate or mean arterial blood pressure of more than 20% of the baseline value after skin incision then it will be considered asblock failure and these patients will be excluded from the study. 1-2ug/kg intravenous fentanyl will be given to failed block. At the end of surgery,residual neuromuscular block will be antagonized with IV neostigmine 0.05 mg/kg and atropine 0.02mg/kg. All patients will receive 15mg/kg paracetamol IV every 6 hours.

Postoperative

1. The postoperative pain assessment in the PACU and the wardwill be performed using a (FLACC score)(APPENDIX 1)(10).Patients will be assessed immediately postoperatively and then at 1st, 4th, 8th, 12th , 24 hour post-operatively.Patients with pain score more than 3\10 ,Pethidine I.V will be given as rescue analgesic (1 mg/kg) when needed.The time to first request of postoperative analgesic is defined as( the time interval from LA injection to first dose of pethidine adminstration) will be recorded. The total amount of pethidine in the first postoperative 24 hours will be calculated in both groups.
2. Block related complications will be recorded such as failed block, local anaesthetic toxicity, vascular puncture, paresthesia.

Measurement tools

1. Patients demographic data will be collected; age, gender, height,weight , type and duration of surgery
2. Block time duration, Surgical procedure , duration and Axillary block performance time.
3. Intraoperative haemodynamic (Heart rate ,systolic and diastolic blood pressure)pre-induction , post-intubation , post-block , immediate post skin incision , every 15 minutes.
4. Postoperative pain assessments using(FLACC score)at at 0 point 1hr, 4hr, 8hr ,12 hr, and at 24 hr
5. Time to first request of rescue postoperative analgesic
6. Total opioid consumption in 24h postoperative
7. Tourniquet whether used or not and if used time and pressure will be recorded

ELIGIBILITY:
Inclusion Criteria:

1. Gender both males and females
2. ASA ClassI-II
3. Age 4-14 years
4. Patients under going upper limb orthopaedic surgery in the hand, wrist, and elbow distal to the cubital fossa

Exclusion Criteria:

1. Parent refusal.
2. Patients with apparent infection at site of needle insertion.
3. Patients with any coagulation disorder(Platelets ≤ 50,000 and/or INR> 1.5)
4. Patients with known neuropathy or brachial plexus injury.
5. Patient with known sensitivity to local anesthetic drugs

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-07-26 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Time to first request of opioid analgesia | it will be measured in the first 24 hours postoperative
  Time to first request of opioid analgesia will be"the time interval between LA injection and the first request to postoperative analgesia (first dose of pethidine adminstration)" (minutes)

SECONDARY OUTCOMES:
Total opioid consumption 24 hours postoperative | It will be measured in the first 24 hours postoperative
  Total opioid consumption will be consumed in the first 24 hours postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed nabih, lecturer, Principal Investigator — Anesthesia department , Cairo university
Locations (1):
- Kasr Alainy, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No